CLINICAL TRIAL: NCT02480205
Title: A Pilot Study of Synchronized and Non-invasive Ventilation ("NeuroPAP") in Preterm Newborns
Acronym: NeuroPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Collaborators: Maquet Cardiovascular (Industry)
Responsible Party: Principal Investigator, Dr Guillaume Emeriaud, MD, PhD, St. Justine's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUSJ-4083
Record Dates: First submitted 2015-05-26; First posted 2015-06-24 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Respiratory Failure
Keywords: CPAP; NIV; NIPPV; Edi
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NeuroBox to deliver the NeuroPAP (Experimental)
  Interventions: Device: NeuroBox to deliver the NeuroPAP

INTERVENTIONS:
Device: NeuroBox to deliver the NeuroPAP — The patients will be studied during the following conditions:
  * On conventional NIPPV device with the clinically prescribed settings (30 min)
  * With NeuroPAP and no change of Pmin (=peep) (60 min)
  * With NeuroPAP and adjusted Pmin (decreased by 2 cmH2O) (60 min)
  * During CPAP delivered with NeuroPAP device (15 min)
  * Again with original NIPPV device and settings for 30 minutes

SUMMARY:
There is currently a consensus that non-invasive ventilation (NIV) in preterm infants is preferred over intubation. There are two ways of delivering NIV in preterm infants, nasal continuous positive airway pressure (CPAP) or nasal intermittent positive pressure ventilation (NIPPV), where ventilator inflations are delivered intermittently over a fixed end-expiratory pressure. The synchronization in conventional mode is very difficult to obtain in premature infants. In all ventilation modes PEEP (end-expiratory pressure) is fixed. Considering that preterm infants are more likely to develop atelectasis, an active and ongoing management of the PEEP is very important to prevent de-recruitment.

A new respiratory support system (NeuroPAP) was developed to address these issues (synchronization problems and control the PEEP). It uses the electrical activity of the diaphragm (EDI) to control the ventilator assist continuously, both during inspiration (principle of NAVA mode) and also during expiration (based on tonic Edi level).

DETAILED DESCRIPTION:
The mode NeuroPAP will work with the continuous Edi-level and deliver pressures according to the Edi-signal x set NeuroPAP-level, over the whole breath (inspiration and expiration). The NeuroPAP will work between two pressure levels set by the user and named higher Pressure limit (Plimit) and minimum Pressure (Pmin).

A safety upper pressure limit (UPL) will also be set. A backup ventilation will be possible.

A specific gastric tube equipped with an array of microelectrodes (Edi catheter, Maquet, Solna, Sweden) will be installed after inclusion, by the same oral or nasal route as the tube previously in place. Patients will then be ventilated in the 5 aforementioned conditions:

* On conventional NIPPV device on clinical settings for a 30 minute period. The investigators will note the mean airway pressure being delivered with the clinical settings and the resulting peak Edi, as well as neural respiratory rate, tonic Edi, Fraction of inspired oxygen (FiO2), and Oxygen saturation by pulse oximetry (SpO2).
* With NeuroPAP without modification of Pmin (=peep). The exchange of the nasal interface may be necessary, depending on the original interface. FiO2 will initially be the same as previously set in conventional NIPPV. The Pmin will initially be set at the level of PEEP used during conventional NIPPV. A titration maneuver will be conducted to identify the optimal NeuroPAP level. The infant will be ventilated for one hour. Clinical adjustments in pressures and FiO2 are permitted. Safety termination will be established.
* NeuroPAP with adjusted Pmin: the Pmin in NeuroPAP will be reduced by 2 cm H2O, with the same NeuroPAP level. The patients will be ventilated for one hour.
* CPAP delivery with NeuroPAP device: the device will be switched to CPAP mode, for a 15 minute period
* A second 30 minutes period of the conventional NIPPV will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants, >26 0/7 and < 34 weeks GA, at least 3 days old and younger than 1 month,
* on NIPPV with settings in the range : Maximal inspiratory pressure (total, including PEEP) < 20 cmH2O, and PEEP : 5-7 cmH2O,
* with FiO2 <40%, and stable.

Exclusion Criteria:

* Suspected or proven pneumothorax
* Patient on high-flow nasal cannula or nasal continuous positive airway pressure (nCPAP)
* Infants with severe recurring apnea
* Recent worsening of respiratory status with increase work of breathing, recent increase in FiO2, or linked with a suspected sepsis
* Contraindications to the placement of a new nasogastric tube (e.g. severe coagulation disorder, malformation or recent surgery in cervical, nasopharyngeal or esophageal regions)
* Hemodynamic instability requiring inotropes.
* Severe respiratory instability requiring imminent intubation according to the attending physician, or FiO2 > 45%, or PaCO2 > 65 mmHg on blood gas in the last hour.
* Patient for whom a limitation of life support treatments is discussed or decided.
* Refusal by the treating physician.

Ages: 3 Days to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2015-08; Primary Completion 2017-01-30 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
Time effectively spent with NeuroPAP mode activated during the NeuroPAP period | up to 30 minutes after reinstitution of the conventional NIPPV
  Percentage
Number of interruption of NeuroPAP during the NeuroPAP period | up to 30 minutes after reinstitution of the conventional NIPPV
  Number of interruption per patients
Change in respiratory rates between standard NIV andNeuroPAP | up to 30 minutes after reinstitution of the conventional NIPPV
  % of change
Change in cardiac rates between standard NIV andNeuroPAP | up to 30 minutes after reinstitution of the conventional NIPPV
  % of change
Change in blood pressure between standard NIV andNeuroPAP | up to 30 minutes after reinstitution of the conventional NIPPV
  % of change
Change in SpO2 between standard NIV andNeuroPAP | up to 30 minutes after reinstitution of the conventional NIPPV
  % of change
Change in TcPCO2 between standard NIV andNeuroPAP | up to 30 minutes after reinstitution of the conventional NIPPV
  % of change

SECONDARY OUTCOMES:
Time spent in asynchrony between standard NIV and NeuroPAP | up to 30 minutes after reinstitution of the conventional NIPPV
  % of time
Change in trigger delays (ms) between standard NIV andNeuroPAP | up to 30 minutes after reinstitution of the conventional NIPPV
Change in non assisted breaths (wasted efforts) between standard NIV andNeuroPAP | up to 30 minutes after reinstitution of the conventional NIPPV
  % of change
Change in autotriggered breaths between standard NIV and NeuroPAP | up to 30 minutes after reinstitution of the conventional NIPPV
  Percentage
Change in Mean Airway pressure (cmH2O) between standard NIV and NeuroPAP | up to 30 minutes after reinstitution of the conventional NIPPV
Change in End expiratory pressure (PEEP, cmH2O) between standard NIV and NeuroPAP | up to 30 minutes after reinstitution of the conventional NIPPV
Change in Mean Electrical activity of diaphragm (Edi, mcV) between standard NIV and NeuroPAP | up to 30 minutes after reinstitution of the conventional NIPPV
Change in Peak Electrical activity of diaphragm (Edi, mcV) between standard NIV and NeuroPAP | up to 30 minutes after reinstitution of the conventional NIPPV
Change in Tonic Electrical activity of diaphragm (Edi, mcV) between standard NIV and NeuroPAP | up to 30 minutes after reinstitution of the conventional NIPPV

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Emeriaud, MD, PhD, Principal Investigator — St. Justine's Hospital; Gregory Lodygensky, MD, PhD, Principal Investigator — St. Justine's Hospital; Jennifer Beck, PhD, Principal Investigator — Li Ka Shing Knowledge Institute. St. Michael's Hospital; Christer Sinderby, PhD, Principal Investigator — Li Ka Shing Knowledge Institute. St. Michael's Hospital
Locations (1):
- St. Justine's Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Rochon ME, Lodygensky G, Tabone L, Essouri S, Morneau S, Sinderby C, Beck J, Emeriaud G. Continuous neurally adjusted ventilation: a feasibility study in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2020 Nov;105(6):640-645. doi: 10.1136/archdischild-2019-318660. Epub 2020 Apr 8. PMID 32269148